CLINICAL TRIAL: NCT03922971
Title: Post-Endoscopic Infection Rate Notifications to Improve the Delivery of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Medivators Cantel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00203304
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-02

CONDITIONS: Infection
Keywords: colonoscopy; EGD; endoscopy; ASC; outpatient; infection; Endoscopic procedures
MeSH Terms: conditions — Infections | interventions — Benchmarking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- National comparison (Other): Ability to view center's rate compared with all others
  Interventions: Other: Option 1: National comparison
- National comparison with benchmarking (Other): Ability to view center's rate compared with the others with a similar patient comorbidity profile and in addition to viewing option 1
  Interventions: Other: Option 2: National comparison with benchmarking

INTERVENTIONS:
Other: Option 1: National comparison — Ability to view center's rate compared with all others.
  Arms: National comparison
Other: Option 2: National comparison with benchmarking — Ability to view center's rate compared with the others with a similar patient comorbidity profile and in addition to viewing option 1.
  Arms: National comparison with benchmarking

SUMMARY:
This project will notify centers of center's post-endoscopic infection rates and evaluate the effectiveness of this notification system to decrease infection rates. The investigators aim to notify centers of the number of patients and center's risk-adjusted rates of hospitalizations for infections after colonoscopy and esophagogastroduodenoscopy (EGD) procedures performed between January 2015 and September 2018. The investigators will randomize centers to two notification groups: (1) Ability to view center's rate compared with all other centers (ASCs and outpatient centers notified and compared separately) or (2) Ability to view center's rate compared with the other centers with a similar patient comorbidity profile and in addition to viewing option 1. Facilities will answer questions about center's infection control practices. The investigators hypothesize that centers with high rates of post-procedural infections will (1) be more likely to report that the center took action to investigate the center's infection control practices after the first notification and (2) observe a decrease in infections after the notification. The investigators anticipate that centers with high rates of post-procedural infections that are randomized to group 2 will have greater change. The investigators anticipate no change in rates of infection in the facilities that had zero or very low (n=1) event rates.

ELIGIBILITY:
Inclusion Criteria:

* Facilities that bill to fee for service Medicare for gastrointestinal endoscopy

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in the infection rate among centers with elevated infection rates | Baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hutfless, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No